CLINICAL TRIAL: NCT00948259
Title: Phase IIa 20 Week Double-blind, Placebo-controlled, Randomized, Escalating Dose Study to Evaluate the Safety and Tolerability of Four Oral Doses of NP031112, a Novel GSK3 Inhibitor, in Mild to Moderate Alzheimer's Disease Patients With Stable Anticholinesterasic Treatment.
Brief Title: Safety Study of a Glycogen Synthase Kinase 3 (GSK3) Inhibitor in Patients With Alzheimer´s Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Noscira SA (Industry)
Responsible Party: Dr. Teodoro del Ser /Medical Director, Noscira SA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP031112-08B03 (CR080901)
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Alzheimer´s Disease
Keywords: safety; GSK inhibitor; Alzheimer
MeSH Terms: interventions — tideglusib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NP031112 (Experimental): Patients will receive 400 mg of NP031112 for 4 weeks, if tolerated, they will receive 600 mg for 4 additional weeks. Patients that tolerate this dose will receive 800 mg for 6 weeks and the patients that tolerate this will escalate to 1000 mg for an additional 6 weeks. Patients that are not eligible for dose escalation will remain on the tolerated dose for the remainder of the study.
  Interventions: Drug: NP031112
- Placebo (Placebo Comparator): Patients will receive 400 mg for 4 weeks, if tolerated, they will receive 600 mg for 4 additional weeks. Patients that tolerate this will receive 800 mg for 6 weeks and the patients that tolerate this will escalate to 1000 mg for an additional 6 weeks. Patients that are not eligible for escalation will remain on the tolerated dose for the remainder of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NP031112 — unidose sachets containing dry powder for oral suspension, once daily dosing 400 mg (4 to 20 weeks), 600 mg(4 to 16 weeks),800 mg (6 to 12 weeks), 1000 mg (6 weeks)
  Other Names: tideglusib; NP12
  Arms: NP031112
Drug: Placebo — unidose sachets containing dry powder for oral suspension, once daily dosing 400 mg (4 to 20 weeks), 600 mg(4 to 16 weeks),800 mg (6 to 12 weeks), 1000 mg (6 weeks)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if 4 escalating doses during 20 weeks of NP031112 are safe and tolerated in patients with Alzheimer´s disease.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women (non-childbearing potential) with a diagnosis of probable Alzheimer's disease according to the NINCDS-ADRDA clinical criteria.
2. Age 60 - 85 years (patients over 85 years could be included after a previous assessment by the investigator and in agreement with the sponsor)
3. MRI or CT-scan assessment within 12 months before baseline corroborating the clinical diagnosis (diffuse brain atrophy predominating in medial temporal regions) and excluding other potential causes of dementia, especially cerebrovascular lesions (see exclusion criteria, number 3).
4. Mild to moderate stage of Alzheimer's disease according to MMSE 16-26.
5. Modified Hachinski ischemic score equal to or below 4.
6. Geriatric Depression Scale below or equal 7.
7. Female patients must be either surgically sterilized or at least 1 year postmenopausal (confirmed by FSH >20, for women not surgically sterilized).
8. A caregiver/nurse is available and is living in the same household, or interacts with the patient to assure the correct preparation and administration of the study drug to the patient.
9. Patients living at home or old people's home.
10. General health status acceptable for a participation in a 6 months clinical trial.
11. Ability to swallow 100 -150 ml of water suspension.
12. No daily-regular/chronic intake of medications acting on central nervous system, immunosuppressants, steroids or non-steroid anti-inflammatory agents except the following allowed treatments:

    * SSRIs as antidepressants if they are administered at a stable and well tolerated dose for two months prior to baseline evaluation
    * the following drugs at a stable and well tolerated dose to symptomatic treatment of mild behavioral disorder, sleep onset-insomnia or mild depressive mood:

      * Risperidon max 1mg/day
      * Quetiapin max 25mg/day
      * Zolpidem max 10mg in the evening
      * Lorazepam max 1mg/day
      * Triazolam max 0,25mg/day
      * Alprazolam max 1mg/day
      * Mirtazapin max 30mg/day
    * Hydromorphon max 4mg/day
    * Levodopa max 50mg t.i.d as treatment of an age-associated extrapyramidal syndrome or restless-legs-syndrome
    * Acetylsalicylic acid max 100mg/day as antiplatelet agent.
    * Non-steroid anti-rheumatics as concomitant medication taken per request
13. No history of treatment with Warfarin, Digitoxin or Coumarin (including its derivatives) within 1 month prior to baseline. Chronic treatment with heparin s.c. as anticoagulant or digoxin for the treatment of heart disease are allowed.
14. Other drugs metabolized by the CYP3A4 with wide therapeutic window are permitted if their dose and regimen are stable and well tolerated for at least 1 month prior to baseline.
15. Stable pharmacological treatment of any other chronic condition for at least one month prior to screening.
16. Treatment with a stable and well tolerated dose of one of the approved Acetylcholinesterase-Inhibitors (Donepezil, Galantamine or Rivastigmine) for at least 2 months prior to baseline evaluations. Dosage of Acetylcholine-esterase inhibitors should not be increased during the ongoing study.
17. No history of treatment with Memantine within 3 months prior to baseline evaluation. Patients with a stable and well tolerated dose of Memantine are not allowed to be included in the study.
18. Signed informed consent by patient prior to the initiation of any study specific procedure

Exclusion Criteria:

1. Failure to perform screening or baseline examinations.
2. Hospitalization or change of chronic concomitant medication within 1 month prior to screening period.
3. Clinical, laboratory or neuroimaging findings consistent with:

   * other primary degenerative dementia, (dementia with Lewy bodies, frontotemporal dementia, Huntington's disease, Jacob-Creutzfeld Disease, Down's syndrome, etc)
   * other neurodegenerative condition (Parkinson's disease, amyotrophic lateral sclerosis, etc.)
   * cerebrovascular disease (major infarct, one strategic or multiple lacunar infarcts, extensive white matter lesions)
   * other central nervous system diseases (severe head trauma, tumors, subdural haematoma or other space occupying processes, etc.)
   * seizure disorder
   * other infectious, metabolic or systemic diseases affecting central nervous system (syphilis, present hypothyroidism, present vitamin B12 or folate deficiency, serum electrolytes out of normal range, juvenile onset diabetes mellitus, etc.)
4. A current DSM-IV diagnosis of active major depression, schizophrenia or bipolar disorder.
5. Clinically significant, advanced or unstable disease that may interfere with evaluations that may bias the assessment of the clinical or mental status of the patient or put the patient at special risk, such as:

   * chronic liver disease, liver function test (LFT) abnormalities or other signs of hepatic insufficiency
   * respiratory insufficiency
   * renal insufficiency (serum creatinine >2mg/dl and creatinine clearance ≤ 60 mL/min according to Cockgroft-Gault formula).
   * heart disease (myocardial infarction, unstable angina, heart failure, cardiomyopathy within 6 months before screening)
   * bradycardia (heart beat <50/min.) or tachycardia (heart beat >95/min.)
   * hypertension or hypotension if not well controlled or unstable for > 2 months prior to baseline.
   * AV block (type II / Mobitz II and type III), congenital long QT syndrome, sinus node dysfunction or prolonged QTcB-interval (males >450 and females >470 msec)
   * uncontrolled diabetes
   * malignant tumors within the last 5 years except skin malignancies (other than melanoma) or indolent prostate cancer
   * metastases
6. Disability that may prevent the subject from completing all study requirements (e.g., blindness, deafness, severe language difficulty, etc.)
7. Women who are fertile and of child bearing potential.
8. Anticoagulant treatment with heparin i.v.
9. Chronic drug intake of:

   * drugs metabolized by the CYP3A4 with narrow therapeutic window (i.e. warfarin, digitoxin, …).
   * antidepressants, benzodiazepines, neuroleptics or sedatives except those defined as allowed in the inclusion criterion number 12
   * proton-pump inhibitors
   * antiepileptics
   * anticholinergics
   * nootropics
   * centrally active anti-hypertensive drugs (clonidine, alpha-methyl dopa, guanidine, guanfacine, …)
   * opioid containing analgesics
   * non-steroid anti-inflammatory agents (except taken as concomitant medication per request as defined in the inclusion criterion number 12), cortico-steroids or immunosuppressants
   * memantine, lithium or other inhibitor of GSK3 enzyme
10. Suspected or known drug or alcohol abuse.
11. Suspected or known allergy to any components of the study treatments.
12. Enrolment in another investigational study or intake of investigational drug within the previous 3 months.
13. Any condition which in the opinion of the investigator makes the patient unsuitable for inclusion.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Incidence rates and severity of clinical adverse events and lab abnormalities for each dose level and placebo | 20 weeks

SECONDARY OUTCOMES:
Effect of treatment with four doses of NP031112 on cognition and depressive mood | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Klaus-Christian Steinwachs, MD, Principal Investigator — Studienzentrum PD Dr. Steinwachs; Manfred Windisch, Ph.D., Study Director — JSW Life Sciences GmbH
Locations (3):
- Germany (3):
  - Pharmacologische Studiecentrum Chemnitz, Chemnitz
  - Arzneimittelforschung Leipzig GmbH, Leipzig
  - Studienzentrum PD Dr. Steinwachs, Nuremberg